CLINICAL TRIAL: NCT06959277
Title: Balance4Mobility: Effects of Walkasins Use on Clinical Outcomes of Gait and Balance Function in Individuals With Peripheral Neuropathy and Balance Problems - A Randomized Control Trial
Brief Title: Balance4Mobility: Effects of Walkasins Use in Individuals With Peripheral Neuropathy and Balance Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RxFunction Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0010
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Neuropathies; Peripheral Neuropathy Due to Chemotherapy; Peripheral Neuropathy With Type 2 Diabetes; Balance Control in Elderly; Gait Disorders
Keywords: Walkasins; Peripheral Neuropathy; Balance Problems
MeSH Terms: conditions — Peripheral Nervous System Diseases; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Control group participants will receive Walkasins after six months of taking part in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Walkasins User Group (Experimental): Participants randomized to the user group will receive Walkasins, consisting of two parts for each leg: the Haptic Module and the Receptor Sole. They will use the device for one year (52 weeks). In addition, the user group participants will receive the fall prevention information provided to the control group.
  Interventions: Device: Walkasins; Other: Fall Prevention Training
- Control Group (Other): Participants randomized to the control group will receive fall prevention information during the baseline visit. After six months, they will receive Walkasins for use during the final six months of the trial.
  Interventions: Other: Fall Prevention Training

INTERVENTIONS:
Device: Walkasins — Walkasins® is an external, lower limb sensory prosthesis intended to replace part of the nerve function used for detection and signaling of foot pressure sensation during standing and walking activities. Walkasins consist of two parts for each leg: the Haptic Module and the Receptor Sole. The Haptic Module wraps around the lower leg of the user and contains electronics for reading Receptor Sole pressure signals, a microprocessor, and four vibrating motors that provide gentle tactile sensory cues to the front, back, medial, and lateral surfaces of the user's leg. These cues reflect real-time foot pressure information at a location above the ankle where skin sensation is still present.
  Arms: Walkasins User Group
Other: Fall Prevention Training — Participants will watch "6 Steps to Prevent a Fall," a short (2 minute) educational video from the National Council on Aging, which describes simple steps to reduce fall risk. To improve their access to the education provided, participants will also receive three handouts, produced by the Center for Disease Control and Prevention (CDC) STEADI initiative (Stopping Elderly Accidents, Deaths, and Injuries), to review after the study visit. The STEADI Initiative is a coordinated approach for healthcare providers to implement the American and British Geriatrics Societies' Clinical Practice Guideline for fall prevention (https://www.cdc.gov/steadi/index.html).

SUMMARY:
The goal of this clinical trial is to is to test whether Walkasins can help people with peripheral neuropathy maintain their balance better. The main question it aims to answer is whether participants who use Walkasins on an everyday basis over a six-month period will report better awareness of their foot placement on the ground.

Researchers will compare Walkasins users to a control group of participants who are not using Walkasins to see if the device improves the users' performance on some standing and walking tests. Control group participants will get Walkasins after six months of being in the study.

During the study participants will be asked to do the following:

* Answer questions about their medical history and balance.
* Do some standing and walking tests. Some of the tests will be timed.
* Attend study visits and participate in study phone calls.
* Keep track of any falls and notify study staff if they fall.
* Wear the Walkasins device on a regular basis.

DETAILED DESCRIPTION:
A randomized cross-over study of short-term, in-clinic effects of Walkasins use, conducted at the Minneapolis Veterans Affairs Medical Center (VAMC) and published in PLOS ONE, found clinically meaningful and statistically significant improvements in gait speed and functional balance in patients with SPN using Walkasins. The authors stated that "findings suggest new sensory balance cues provided to the lower limb can modulate the activity of relevant nerve afferents and become integrated into sensorimotor control of balance and gait."

In 2020 a multi-site clinical trial of the long-term effects of daily Walkasins use (walk2Wellness, ClinicalTrials.gov #NCT03538756) was published in Frontiers in Aging Neuroscience. After 10 weeks of Walkasins use, this long-term study demonstrated clinically meaningful improvements in Functional Gait Assessment (FGA) and gait speed, which is associated with a lower fall risk. The authors concluded that "a wearable sensory prosthesis may provide a new way to treat gait and balance problems and manage falls in high fall-risk patients with PN."

Most recently, an analysis of data from 26 weeks of Walkasins use in the walk2Wellness trial showed that "participants who reported falls over 6 months prior to the study had a 43% decrease in fall rate during the study as compared to self-report 6-month pre-study (11.8 vs. 6.7 falls/1000 patient days, respectively, p <0.004), similar to the 46% decrease reported after 10 weeks of use."

The present study involves an assessment of Walkasins through a randomized, controlled trial with a primary endpoint of 26 weeks. Furthermore, this study will enroll only individuals 55 and older with a goal of including participants that reflect the Medicare population to support payer reimbursement for Walkasins.

The objectives of this study are as follows:

* Reflect real-world use of Walkasins in a Medicare-representative population who have sensory peripheral neuropathy and associated gait and balance problems and who would be eligible for a prescription to use the device.
* Investigate the impact of Walkasins use on relevant clinical outcomes associated with gait and physical function.
* Demonstrate based on patient reporting that Walkasins improves awareness of foot placement on the ground indicating partial replacement of plantar mechanoreceptor function, lost due to peripheral neuropathy.
* Investigate whether plantar monofilament testing at levels <10g (5.07, LOPS) are associated with gait and balance issues. Is there a Loss Of Balance Sensation (LOBS) threshold that is <10g? The monofilament test protocol should include plantar sites across the foot since differences in anteroposterior and/or mediolateral sensitivity may cause balance issues.
* Compare the rate of injurious falls between a group of Walkasins users and non-users over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent for him or herself
* Age 55 and older, male or female
* Able to complete all functional outcome measures without the use of an assistive device
* Clinical diagnosis of peripheral neuropathy prior to participating in the study as documented in the participant's medical record or by physician's note. Individuals with chemo-induced peripheral neuropathy must be at least one-year post-chemotherapy, indicating that their PN has become a chronic condition.
* Self-reported gait and balance problems
* Foot size that allows the Walkasins to function appropriately
* Willing to use the Walkasins device as recommended

Exclusion Criteria:

* Ability to stand on one leg for at least 30 seconds (If the person can stand for at least 30 seconds, he/she is excluded because his/her balance is likely not impaired enough to benefit from Walkasins.)
* Self-reported acute thrombophlebitis, including deep vein thrombosis
* Self-reported severe peripheral vascular disease
* Untreated lymphedema
* Untreated lesion of any kind, swelling, infection, inflamed area of skin or eruptions on the lower leg near product use
* Self-reported, untreated fractures in the foot and ankle
* Other neurological or musculoskeletal conditions that moderately or severely impact walking
* Use of ankle-foot orthosis for ambulation that prevents donning of Walkasins
* Weight of more than 300 pounds
* Inability to perceive vibration from Walkasins Haptic Module

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment (FGA) | Baseline, Week 10, Week 26, Week 36 (Control Group), and Week 52
  The Functional Gait Assessment (FGA) is a 10-item scale that measures postural stability while individuals perform walking tasks that are scored from 0 to 3 (3 = normal, 2 = mild impairment, 1 = moderate impairment, 0 = severe impairment). Scores range from a minimum of 0 to a maximum of 30. Higher scores indicate better postural stability.
Patient-Specific Functional Scale (PSFS) | Baseline, Week 5, Week 10, Week 18, Week 26, Week 31, Week 36, Week 41, Week 46, and Week 52
  The PSFS asks patients to define up to five specific tasks that they have difficulty with or are unable to perform because of their physical injury or disability. Some research studies adapt the PSFS by asking participants to list three tasks rather than five, which is the plan for this study. The patients then rate their difficulty in performing those tasks on a scale of 0 to 10 with 0 meaning "unable to perform activity" to 10 meaning "able to perform activity at the same level as before injury or problem." The ratings for the three activities are averaged. Higher scores indicate greater ability to perform the activity.
PROMIS® PROWalk | Baseline, Week 5, Week 10, Week 18, Week 26, Week 31, Week 36, Week 41, Week 46, and Week 52
  Eight items that have the most relevance for measuring change in individuals who have received Walkasins were selected from the 165 items comprising the PROMIS Item Bank v2.0 - Physical Function. Specifically, the selected items measure an individual's ability to perform various activities that involve upright mobility (balance, standing, and walking). Participants rate the eight items on a scale of 1 to 5; the raw scores are converted to T-scores for comparison to national norms.

SECONDARY OUTCOMES:
10-Meter Walk Test | Baseline, Week 10, Week 26, Week 36 (Control Group), and Week 52
  Gait speed will be measured through the 10-Meter Walk Test, timing only the middle 6 meters to allow for acceleration and deceleration. Participants will be instructed to walk at normal speed. Higher numbers indicate faster speeds (i.e., more meters per second).
Four-Stage Balance Test | Baseline, Week 10, Week 26, Week 36 (Control Group), and Week 52
  The 4-Stage Balance Test is part of the Centers for Disease Control's recommended test protocol for balance function. It includes four gradually more challenging postures the subject is exposed to: (1) Stand with feet side by side. (2) Stand with feet in semi-tandem stance. (3) Stand with feet in tandem stance. (4) Stand on one leg. Participants pass each level if they can hold the stance for 10 seconds and then move on to the next stance. If they cannot hold the stance, the test ends. Higher times indicate better balance than lower times.
Modified Multidirectional Reach Test | Baseline, Week 10, Week 26, Week 36 (Control Group), Week 52
  The Multidirectional Reach Test is a quick screening tool for fall risk to indirectly measure the limits of stability. The participant outstretches his/her arm to shoulder height next to a yardstick mounted on the wall; then he/she reaches as far as possible in the instructed direction without taking a step. The test administrator records the start and end position of the index finger of the outstretched hand, and the difference represents the total reach for that direction. Higher differences indicate better stability.
  The Modified Multidirectional Reach Test used in this clinical trial will include only forward and backwards reaching that is completed and recorded with eyes closed. It will omit the left and right reaches.
Single Leg Stance Test | Baseline, Week 26
  The Single Leg Stance Test (also called the unipedal stance test) "is a simple test for measuring static aspects of balance." It "is related to conditions such as peripheral neuropathy and intermittent claudication" and "is also associated with an increased risk for falls" (Spring et al., 2007) Participants stand unassisted on one leg with their hands on their hips. Timing begins when they lift one leg off the floor and ends when it touches the ground or the standing leg or an arm leaves the hips
Timed Up and Go (TUG) and Timed Up and Go Cognitive/Dual Task (TUG-COG) | Baseline, Week 10, Week 26, Week 36 (Control Group), Week 52
  The Timed Up and Go Test is part of the Centers for Disease Control (CDC)-recommended STEADI test protocol for balance function. From a seated position in a standard armchair, the participant is asked to stand up from the chair, walk to a line on the floor 10 feet away at normal pace, turn, walk back to the chair at normal pace, and sit down again. The tester records the time taken from the command "Go" until the subject sits down again. Lower times indicate better/faster performance.
  The TUG-Cog is performed as described above; in addition, the participant is asked to count backwards by threes from a randomly selected number between 20 and 100. Lower times indicate better/faster performance.
Activities-specific Balance Confidence Scale 6 (ABC-6) | Baseline, Week 5, Week 10, Week 18, Week 26, Week 31, Week 36, Week 41, Week 46, and Week 52
  Powell and Myers developed the 16-item Activities-specific Balance Confidence (ABC) Scale to detect levels of balance confidence in older adults. Schepens et al. (2009) validated a 6-item version of the ABC, using the six most challenging activities from the 16-item scale. The six tasks are rated on a scale of 0 to 100; a score of 0 indicates no confidence and a score of 100 indicates complete confidence when performing the task. The overall score is calculated by adding the individual items then dividing by the total number of items (6). The higher the score, the greater the person's balance confidence; thus, higher scores indicate that subjects are more confident of their balance.
EuroQol HRQoL (EQ-5D-5L) | Baseline, Week 10, Week 26, Week 36, and Week 52
  The EQ-5D-5L consists of five questions, one each on "mobility," "self-care," "usual activities," "pain / discomfort," and "anxiety / depression." Participants rate themselves according to statements reflecting five levels ranging from no problems with the activity or construct to inability to perform the activity or having an extreme amount of difficulty with the construct.
PROMIS® Scale v2.0 - Pain Intensity 3a and Neuropathic Foot Pain Rating | Baseline, Week 10, Week 26, Week 36, Week 52
  The PROMIS Pain Intensity assessment measures "how much a person hurts" (https://www.healthmeasures.net/images/PROMIS/manuals/PROMIS_Pain_Intensity_Scoring_Manual.pdf). The three questions are not disease specific. Two items address pain experienced in the past seven days; the other, pain at present. In addition, we will ask participants to rate the neuropathic pain in their feet on scale of 0-10 (0 = No Pain, 10 = Worst Pain Imaginable).
Rapid Assessment of Physical Activity (RAPA) and Telephone Assessment of Physical Activity (TAPA) | Baseline, Week 10, Week 18, Week 26, Week 36, and Week 52
  The Rapid Assessment of Physical Activity (RAPA) is a measure of physical activity, designed for use with older adults. The researchers will administer the RAPA during in-person visits and the TAPA, a telephone-based assessment of physical activity based on the RAPA, during the Weeks 18 and 36 telephone visits. The assessments consist of seven questions on light, moderate, and vigorous physical (aerobic) activities to which the participants respond "yes" or "no," depending on whether or not the question is true of them. Scoring is based on the number of the item to which the participants report the highest positive response (e.g., if the participant answered "Yes" to question 4 and "No" to 5, 6, and 7, then "4" is the participant's score). Higher scores indicate more physical activity. The final two items address strength and flexibility and are scored separately.
Walkasins Experience Survey | Baseline, Week 10, Week 26, Week 36 (Control Group), and Week 52
  At the follow-up visits, the study team will ask the participants assigned to the Walkasins user group specific questions about their experience with Walkasins. Control group participants will complete the survey at Weeks 36 and 52.

OTHER OUTCOMES:
Falls Monitoring | Week 5, Week 10, Week 18, Week 26, Week 31, Week 36, Week 41, Week 46, and Week 52
  Participants will report details regarding falls they experience during their enrollment in the study.
Monofilament Test | Baseline, Week 26, and Week 52
  The Centers for Medicare & Medicaid Services (CMS) identifies the monofilament test as the means of diagnosing loss of protective sensation (https://www.cms.gov/medicare-coverage-database/view/ncd.aspx?NCDId=171). To conduct the test, a clinician applies pressure with various sizes of monofilament to selected parts of the foot and asks the participant to indicate when he/she feels the filament. Including catch trials helps to ensure accurate test results. Per CMS, inability to feel a 10-gram monofilament on at least two of five test sites on either foot indicates loss of protective sensation (LOPS).
Vibration Test | Baseline, Week 26, and Week 52
  Vibration is one of several types of sensation encompassed within the somatosensory system, and it is often diminished in individuals with neuropathy. To examine vibration sense, a clinician applies a low-frequency (128 Hz) tuning fork to bony prominences and asks the participant (with closed eyes) to report when the vibration starts and stops. For this study, site personnel will employ the Rydel-Seiffer tuning fork, which provides a more quantitative assessment of vibratory sensation ranging from 2 to 8.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Oddsson, PhD, Study Director — RxFunction Inc.
Locations (6):
- United States (6):
  - OrthoArizona--Mesa Arbor Avenue, Mesa, Arizona
  - Marcus Institute for Aging Research, Hebrew SeniorLife, Boston, Massachusetts
  - Fairview Frontiers, Saint Paul, Minnesota
  - Dent Neurologic Institute, Amherst, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor will make a determination on data sharing prior to publication of the results.

REFERENCES:
- [Background] Hsu CL, Manor B, Iloputaife I, Oddsson LIE, Lipsitz L. Six month lower-leg mechanical tactile sensory stimulation alters functional network connectivity associated with improved gait in older adults with peripheral neuropathy - A pilot study. Front Aging Neurosci. 2022 Nov 3;14:1027242. doi: 10.3389/fnagi.2022.1027242. eCollection 2022. PMID 36408098
- [Background] Koehler-McNicholas SR, Danzl L, Cataldo AY, Oddsson LIE. Neuromodulation to improve gait and balance function using a sensory neuroprosthesis in people who report insensate feet - A randomized control cross-over study. PLoS One. 2019 Apr 30;14(4):e0216212. doi: 10.1371/journal.pone.0216212. eCollection 2019. PMID 31039180
- [Background] Oddsson LIE, Bisson T, Cohen HS, Iloputaife I, Jacobs L, Kung D, Lipsitz LA, Manor B, McCracken P, Rumsey Y, Wrisley DM, Koehler-McNicholas SR. Extended effects of a wearable sensory prosthesis on gait, balance function and falls after 26 weeks of use in persons with peripheral neuropathy and high fall risk-The walk2Wellness trial. Front Aging Neurosci. 2022 Sep 20;14:931048. doi: 10.3389/fnagi.2022.931048. eCollection 2022. PMID 36204554
- [Background] Oddsson LIE, Bisson T, Cohen HS, Jacobs L, Khoshnoodi M, Kung D, Lipsitz LA, Manor B, McCracken P, Rumsey Y, Wrisley DM, Koehler-McNicholas SR. The Effects of a Wearable Sensory Prosthesis on Gait and Balance Function After 10 Weeks of Use in Persons With Peripheral Neuropathy and High Fall Risk - The walk2Wellness Trial. Front Aging Neurosci. 2020 Nov 9;12:592751. doi: 10.3389/fnagi.2020.592751. eCollection 2020. PMID 33240077
- See also: RxFunction is the manufacturer of Walkasins. The website provides additional information about the device. — https://www.rxfunction.com/